CLINICAL TRIAL: NCT06121076
Title: A Cross-cultural Project of the Tailored EBP-SDM Training Program Empowers Nurses and Midwives in Competency and Performance.
Brief Title: Effects of the Shared-decision Making Training Program
Acronym: SdmEbp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Quyen Thao Nguyen, lecturer, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SdmEbp2023
Record Dates: First submitted 2023-10-23; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Competence
Keywords: shared-decision making; evidence-based practice; midwife

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDM-EBP training (Experimental): the group received SDM combined with EBP training
  Interventions: Other: SDM-EBP training
- control (Other): the group received received SDM without EBP training
  Interventions: Other: SDM-EBP training

INTERVENTIONS:
Other: SDM-EBP training — A 20-hour tailored SDM combined with EBP training program consisting of a seven-hour lecture and a four-hour hands-on practice session.

SUMMARY:
The goal of this intervention study is to test the effectiveness of a training program for hospital-based midwives. The main questions it aims to answer are: •Does SDM combined EBP training improve midwives' SDM and EBP competency? • What are factors related to SDM competency in midwives? Participants will participate in a 20-hour training program, including lectures and hands-on practice sessions. Researchers will compare groups that receive SDM training with or without EBP training to see if there are changes in midwives' SDM and EBP competency.

DETAILED DESCRIPTION:
This study aimed to evaluate the effect of SDM training program, with or without EBP, on the level of midwives' SDM and EBP competency. This randomized controlled trial recruited participants from 18 departments of an obstetrics and gynecology hospital in Vietnam. 72 midwives (36 in each group) and 404 patients were required. Eligible midwives were ones who provided the hands-on care of patients for at least three months, were licensed to practice midwifery, and were willing to participate in the study. Each participating midwife conducted three encounters with real patients who were conveniently selected. Patients at least 18 years old, having SURE test scores less than 4, and willing to participate in the study were invited. Patients requiring emergency medical attention were excluded. The intervention group received a tailored training program that combined SDM with EBP, while the control group received SDM training alone. The outcomes related to SDM (measured by SDM-Q-Doc, SDM-Q-9, DSC, OPTION5, DSAT10, and 4HCS) and EBP (measured by HS-EBP) were evaluated at baseline, Week 2, and/or Week 4.

ELIGIBILITY:
Inclusion Criteria for midwives:

* provide hands-on care to patients for at least three months
* licensed to practice midwifery
* willing to participate in the study.

Inclusion Criteria for patients:

* having SURE test score less than 4 (SURE was a decisional conflict screening tool. A score less than 4 was a positive result for decisional conflict)
* willing to participate in the study

Exclusion Criteria for patients:

* Patients requiring emergency medical attention

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
SDM competency from midwives' perspective | baseline, week 2, week 4
  The SDM competency from a midwife's perspective is defined as the ability perceived by midwives to involve patients in the decision-making process. It is measured using the 9-item Shared Decision-Making Questionnaires for healthcare professionals (SDM-Doc). The questionnaire consists of 9 items, and each item represents a statement that features various aspects of SDM using a 6-point Likert scale from 0 (completely disagree) to 5 (completely agree). A total score ranged from 0~45; higher scores indicate a higher level of SDM competency.
SDM competency from observers' perspective | baseline, week 2, week 4
  The SDM competency, from the observers' perspective, is defined as the efforts of healthcare professionals to involve patients in decision-making from blinded observers. It is measured by the Observing Patient Involvement scale (OPTION5). Each item was scored on a 5-point scale from 0 (no effort) to 4 (exemplary effort). A total score ranged from 0~20, with higher scores and higher levels of the extent to which healthcare providers involved patients in decision-making.
SDM competency from patients' perspective | baseline, week 2, week 4
  The SDM competency from a patient's perspective is defined as the patient's perceived extent to which SDM has taken place in the encounter with midwives. It is measured using the 9-item Shared Decision-Making Questionnaires for patients (SDM-Q-9). The questionnaire consists of 9 items, and each item represents a statement that features various aspects of SDM using a 6-point Likert scale from 0 (completely disagree) to 5 (completely agree). A total score ranged from 0~45; higher scores indicate a higher level of SDM competency.
Decision support skill | baseline, week 2, week 4
  Decision support skill is defined as midwives' competency to support patients during the decision-making process. It is measured from blinded observers using the Decision Support Analysis Tool (DSAT10). DSAT10 has five categories of decision-making status, knowledge of options, values associated with outcomes of options, others' involvement, and next steps plan. Assessing and intervening are differentiated in the scale. Each check item was rated as present (1) or absent (0). Not applicable was used in circumstances when it was not necessary to have met an item. A total score ranged from 0~10, with higher scores for better SDM skills.
Communication skill | baseline, week 2, week 4
  Communication skill is defined as midwives' competency to express verbal and non-verbal behaviors of patient- and relationship-centered communication. It is measured from blinded observers using the Four Habits Coding Scheme. The 4HCS consisted of 23 items with four habits of basic medical interview, including invest in the beginning (6 items), elicit the patient's perspective (3 items), demonstrate empathy (4 items), and invest in the end (10 items). Each item was scored on a 5-point scale from 1 (ineffective) to 5 (highly effective). A total score ranged from 23~115, with higher scores for more effective patient-centered communication in consultations.

SECONDARY OUTCOMES:
Level of EBP competency | baseline, week 2, week 4
  The EBP competency is defined as attitude, knowledge, and skill that is perceived by midwives toward evidence-based practice. It is assessed using the Health Sciences-Evidence Based Practice questionnaire (HS-EBP). The 60-item HS-EBP includes five domains of beliefs-attitudes (12 items), results from scientific research (14 items), development of professional practice (10 items), assessment of results (12 items), and barriers-facilitators (12 items). Each item was rated on a 10-point Likert scale (ranging from 1 to 10), with higher scores indicating a greater degree of agreement.
Decision conflict | baseline, week 2, week 4
  Decision conflict is defined as the degree of conflict experienced by patients when making treatment-related decisions. It is measured by the Decision Conflict scale (DCS). DCS had 16 items and is covered by five subscales, including informed (3 items), values clarity (3 items), social support (3 items), uncertainty (3 items), and effective decision (4 items). Each item was scored on a 5-point Likert scale from 0 (strongly agree) to 4 (strongly disagree). In each subscale, the scores of the items were summed up, divided by the number of items, and multiplied by 25, with a possible score ranging from 0 (no decision conflict) to 100 (extremely high decision conflict). A score below 25 indicated the implementation of the decision, and scores exceeding 37.5 signify decision delay or feeling unsure about implementing their decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-ling Yeh, PhD, Study Director — National Taipei University of Nursing and Health Sciences
Locations (1):
- Obstetric hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No